CLINICAL TRIAL: NCT06628830
Title: Efficacy of a Mobile Phone Application for Early Intervention of Depression and Anxiety in Young College Students
Brief Title: Efficacy of a Mobile Phone App for Depression and Anxiety in College Students
Acronym: VamosJuntxs
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: University of Talca (Other); Universidad de los Andes, Chile (Other); Universidad Austral de Chile (Other); Millennium Nucleus to Improve the Mental Health of Adolescents and Youths (Imhay) NCS2021_081 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fondecyt 1221230
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
Keywords: digital intervention; depression; anxiety; app-based Intervention; university students; well-being; college students; mobile phone app
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention consists of an indicated prevention program delivered through a mobile app. The program will last 6 weeks and includes the following:
  1. Psychoeducation on depression and anxiety
  2. CBT skills training
  3. mood and symptom monitoring and feedback: mood tracker and the application every two weeks of the PHQ-4 and question 9 of the PHQ-9
  4. Chat with a psychologist (on demand)
  5. Optional modules on other related mental health topics (e.g. healthy habits, relaxation, mindfulness)
  Additionally, participants will be able to access additional help resources that include a speed dial button for a suicide prevention hotline and a web link to access contact information for mental health services. Finally, the intervention protocol also includes the eventual referral to face-to-face mental health care if required.
  Interventions: Device: VamosJuntxs App
- Control Group (Active Comparator): Participants in the enhanced control group will receive a web link (https://concienciasaludable.uchile.cl/) with information about places to go to seek mental health care both inside and outside the respective university and psychoeducational material on depression and anxiety
  Interventions: Other: Web Conciencia Saludable

INTERVENTIONS:
Device: VamosJuntxs App — Psychoeducational materials (videos, information and interactive exercises) about depression, anxiety and social support
  Skills training through information and activities based on the principles of cognitive behavioral therapy (cognitive restructuring, behavioral activation, emotional regulation, problem solving and exposure)
  Arms: Intervention Group
Other: Web Conciencia Saludable — mental health psychoeducational campaign (https://concienciasaludable.uchile.cl/)
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a mobile phone application for the early intervention of depression and anxiety among young university students in Chile. The main question it aims to answer is:

- Can a mobile app reduce depressive and anxious symptomatology in college students?

Researchers will compare the intervention arm (mobile app users) to the control group (receives psychoeducational material and mental health care resources) to see if the app leads to significant improvements in depressive and anxious symptoms and well-being.

Participants will:

* Be randomly assigned to either the intervention or control group.
* Use the mobile application, which includes psychoeducational materials, cognitive-behavioral therapy modules, and periodic personalized feedback.
* Complete assessments at baseline, post-intervention, and 3 and 6 months after randomization using online tools such as the PHQ-9 for depressive symptoms and the GAD-7 for anxious symptoms.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 and GAD-7 score between 5 and 14 points
* Have a stable internet connection
* To provide informed consent

Exclusion Criteria:

* High risk of suicide according to C-SSRS
* Currently undergoing psychological, psychiatric and/or psychopharmacological treatment
* Bipolar disorder, psychotic disorder or substance use disorder assessed with the respective modules of the MINI interview.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | 6-weeks post-randomization
  PHQ-9, total score varies between 0 and 27, higher values represent a worse outcome
Anxiety symptoms | 6-weeks post-randomization
  GAD-7, total score varies between 0 and 21, higher values represent a worse outcome

SECONDARY OUTCOMES:
Well-being | 6-weeks post-randomization
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS), total score varies between 7 and 35, higher values represent a better outcome
User Satisfaction | 6-weeks post-randomization
  Ad-hoc satisfaction questionnaire for the intervention group, total score varies between 7 and 28, higher values represent a better outcome and an overall index with values ranging from 1 to 10
Depression symptoms | 3-months post-randomization
  PHQ-9, total score varies between 0 and 27, higher values represent a worse outcome
Anxiety symptoms | 3-months post-randomization
  GAD-7, total score varies between 0 and 21, higher values represent a worse outcome
Well-being | 3-months post-randomization
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS), total score varies between 7 and 35, higher values represent a better outcome
Depression symptoms | 6-months post-randomization
  PHQ-9, total score varies between 0 and 27, higher values represent a worse outcome
Anxiety symptoms | 6-months post-randomization
  GAD-7, total score varies between 0 and 21, higher values represent a worse outcome
Well-being | 6-months post-randomization
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS), total score varies between 7 and 35, higher values represent a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CEMERA, Faculty of Medicine, Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lira D, Caviedes P, Martinez V. Adaptation of a mobile app for early anxiety and depression intervention in university students in Chile: participatory study. BJPsych Int. 2023 May;20(2):37-41. doi: 10.1192/bji.2023.1. PMID 38414999